CLINICAL TRIAL: NCT04718181
Title: Risdiplam - A Phase I, Open-Label, Multi-Period Crossover Study to Investigate the Safety, Food Effect, Bioavailability and Bioequivalence of Oral Doses of Two Different Formulations in Healthy Subjects
Brief Title: Bioavailability and Bioequivalence of Two Risdiplam Tablets in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BP42066
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam; Omeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Cohort A+B: participants will receive, in a five-period crossover way, a single oral dose of risdiplam oral solution 5 mg in fasted state and thereafter risdiplam/F21 or F22 dispersible tablet 5 mg as tablet in fasted and fed states; tablet dispersed in water in fasted and fed states, with a 14-day wash-out period in between the single-dose administrations.
  Cohort C+D: participants will receive, in a two-period fixed sequence design, a single dose of risdiplam/F21 or F22 dispersible tablet 5 mg in fasted state and omeprazole 40 mg once daily for 7 days + a single dose of risdiplam/F21 or F22 dispersible tablet 5 mg in fasted state, on the 7th day of omeprazole. There will be a 14-day wash-out between the two treatment periods.
  Cohort E: participants will receive, in a two-period crossover design, a single oral dose of risdiplam oral solution 5 mg in fasted and fed states, with a 14-day wash-out period in between the single-dose administrations.
  Interventions: Drug: risdiplam; Drug: omeprazole
- Part 2 (optional) (Experimental): Group 1: participants will receive, in four-period crossover design, a single oral dose of risdiplam oral solution 5 mg in both fed and fasted states and the selected dispersible tablet (F21) as swallowed tablet in both fed and fasted states.
  Group 2: participants will receive, in four-period crossover design, a single oral dose of risdiplam oral solution 5 mg in both fed and fasted states and the selected dispersible tablet (F21) as tablet dispersed in water in both fed and fasted states.
  Interventions: Drug: risdiplam
- Part 3 (optional) (Experimental): Group 1: participants will receive, in four-period crossover design, a single oral dose of risdiplam oral solution 5 mg in both fed and fasted states and the selected dispersible tablet (F22) as swallowed tablet in both fed and fasted states.
  Group 2: participants will receive, in four-period crossover design, a single oral dose of risdiplam oral solution 5 mg in both fed and fasted states and the selected dispersible tablet (F22) as tablet dispersed in water in both fed and fasted states.
  Interventions: Drug: risdiplam

INTERVENTIONS:
Drug: risdiplam — Risdiplam will be administered orally at a single dose of 5 mg in different formulations. Dispersible tablet formulations (F21/F22) will be administered as swallowed tablet or as tablet dispersed in water. The powder for constitution to an oral solution will be administered as an oral solution constituted with purified water.
  Other Names: Evrysdi
Drug: omeprazole — Omeprazole will be administered orally as a capsule at a dose of 40 mg per day
  Other Names: Non-investigational medicinal product
  Arms: Part 1

SUMMARY:
The study is a randomized, single oral dose, crossover study in up to three parts to investigate the relative bioavailability and bioequivalence of two different formulations of risdiplam 5 mg (dispersible tablets) versus the current risdiplam oral solution formulation in healthy male and female participants. The effect of food on these two dispersible tablets and the current oral solution will be studied, as well as the effect of omeprazole on the dispersible tablets.

DETAILED DESCRIPTION:
Part 1 of the study is an exploratory comparison of the relative oral bioavailability of the two dispersible tablets versus risdiplam powder for oral solution as the reference. The effect of food on the bioavailability of the two dispersible tablets will be assessed by comparing fed and fasted states in a five-way crossover manner. It will also be assessed whether antacids (omeprazole) have an impact on the bioavailability of the dispersible tablets in a two-way crossover manner. The food effect on the risdiplam oral solution will also be assessed by comparing fed and fasted states in a two-way crossover manner.

In Part 2, based on the data obtained in Part 1 and provided data support further evaluation, a bioequivalence assessment and a food-effect evaluation will be conducted in two groups with the selected dispersible tablet formulation. Each group will randomly receive, in a four-way crossover, a single dose of risdiplam oral solution 5 mg in both fed and fasted states, and a single dose of the selected dispersible tablet in both fed and fasted states.

In Part 3, provided Part 1 data support further evaluation of the second formulation, the second formulation may be assessed for bioequivalence in the same way as described in Part 2.

Enrollment of the same participant in more than one cohort or group will not be permitted regardless of the study part.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) of 18.0 to 32.0 kg/m2
* Male participants, whose partners are women of childbearing potential (WOCBP) or pregnant, must remain abstinent or use adequate contraception methods (both male participant and non-pregnant WOCBP partner) during the treatment period and until 4 months after the last dose of risdiplam or for pregnant female partners during the treatment period and until 28 days after the last dose of risdiplam. Males must refrain from donating sperm during the treatment period and until 4 months after the last dose of risdiplam.
* Willingness and ability to complete all aspects of the study
* A female subject is eligible to participate if she is a woman of non-childbearing potential (WONCBP)

Exclusion Criteria:

* History of any clinically significant gastrointestinal (Gl), renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological, or allergic disease, metabolic disorder, cancer or cirrhosis
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study, including but not limited to the following: Any major illness within 1 month before screening or any febrile illness within 1 week prior to screening and up to first study drug administration
* History or evidence of any medical condition potentially altering the absorption, metabolism, or elimination of drugs
* Surgical history of the GI tract affecting gastric motility or altering the GI tract (with the exception of uncomplicated appendectomy and hernia repair; a cholecystectomy is exclusionary)
* History or presence of clinically significant ECG abnormalities (at Screening only) or cardiovascular disease (e.g., cardiac insufficiency, coronary artery disease, cardiomyopathy, congestive heart failure, family history of congenital long QT syndrome, family history of sudden death)
* History of malignancy in the past 5 years
* Confirmed systolic blood pressure (BP) >140 or <90 mmHg, and diastolic BP >90 or <50 mmHg at Screening only
* Confirmed resting heart rate >100 or <40 beats per minute (bpm) at Screening only
* Clinically significant abnormalities in laboratory test results including hematology, chemistry panel, and urinalysis
* Positive result on human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B virus, or hepatitis C virus (serology) tests at Screening only
* Any suspicion or history of alcohol abuse and/or any history or suspicion of regular consumption/addiction of drugs of abuse within 2 years prior to study drug administration or a positive drug screen test as performed at Screening
* Any consumption of tobacco- or nicotine-containing products from 1 month before Check-in until the end of the study
* Donation of blood or blood products for transfusion over 500 mL within 3 months prior to first study drug administration and for the duration of the study
* Currently enrolled in a clinical study involving another investigational product or in any other type of medical research, or have received the last dose of another investigational product within the last 90 days from clinic check-in (Day -1).
* Use of any prescription (other than hormone replacement therapy) or over-the-counter medications, including herbals and vitamins, within 30 days prior to Check-in
* Any clinically significant history of hypersensitivity or allergic reactions, either spontaneous or following study drug administration, or exposure to food or environmental agents
* History of hypersensitivity to any of the excipients in the formulation of the study drug
* Participants under judicial supervision, guardianship, or curatorship

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Part 1: Plasma Concentration of Risdiplam in Cohorts A and B | Day 1 to Day 7 in Periods 1-5
Part 1: Plasma Concentration of Risdiplam in Fed and Fasted States in Cohort E | Day 1 to Day 7 in Period 1 and Period 2
Part 1: Plasma Concentration of Risdiplam in Cohorts C and D | Period 1: Day 1 to Day 7; Period 2: Day 1 to Day 13
Parts 2 and 3: Plasma Concentration of Risdiplam | Day 1 to Day 11 in Periods 1-4

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events and Serious Adverse Events | Part 1: up to Day 20 in Periods 1-2, up to Day 14 in Periods 3-5; Parts 2 and 3: up to Day 11 in Periods 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Daytona Beach Clinical Rsch Unit, Daytona Beach, Florida
  - QPS- Springfield, Springfield, Missouri
  - Dallas Clinical Research Unit, Dallas, Texas
  - Covance Clinical Research Unit, Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).